CLINICAL TRIAL: NCT00502528
Title: Endothelin Receptor Blockade in Acute ST-elevation Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Irene Lang, PI, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BQ123AMI12/06
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: Infarction; Endothelin; Perfusion
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Infarction | interventions — cyclo(Trp-Asp-Pro-Val-Leu)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): BQ-123
  Interventions: Drug: BQ-123

INTERVENTIONS:
Drug: Placebo — Peri-interventional
  Other Names: sodium salt
  Arms: 1
Drug: BQ-123 — Peri-interventional
  Other Names: Cyclo(-D-Trp-D-Asp-Pro-D-Val-Leu) sodium salt
  Arms: 2

SUMMARY:
Background and Objective: Acute coronary syndrome is characterized by compromised blood flow at the epicardial and microvascular levels. The aim of the present study is to investigate the effect of ET-receptor blockade by BQ-123 on myocardial perfusion and infarct size as an adjunct to PCI-reperfusion therapy in patients with STEMI.

Patients are randomized to receive periinterventional intravenous BQ-123 or placebo.

DETAILED DESCRIPTION:
Background and Objective: Acute coronary syndrome is characterized by compromised blood flow at the epicardial and microvascular levels. We have previously shown that thrombectomy in ST-elevation myocardial infarction (STEMI) accelerates ST-segment resolution, possibly by preventing distal embolization. Therefore, we analyzed the vasoconstrictor concentration of acute coronary thrombi, and found high concentrations of endothelin (ET) which correlated with the magnitude of ST-segment resolution within one hour of percutaneous coronary intervention (PCI). Furthermore, ET-receptor blockade by tezosentan significantly repressed vasoconstriction in an in-vitro model using porcine coronary artery rings incubated with coronary thrombus homogenates extracted from STEMI patients.

The aim of the present study is to investigate the effect of ET-receptor blockade by BQ-123 on myocardial perfusion and infarct size as an adjunct to PCI-reperfusion therapy in patients with STEMI.

Methods: Fifty eligible patients will be randomized to receive periinterventional intravenous BQ-123 or placebo. The primary endpoint of the study will be microvascular function evaluated by cardiac magnetic resonance tomography.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients (defined as: Evidence of ischemic chest pain for >30 minutes within <12 hours and new ST-segment elevation for ≥2 mm in two or more contiguous electrocardiographic leads or in case of a true posterior infarction reciprocal ST-segment depressions in in V1 and V2 >1mm and/or elevated serum creatine phosphokinase or twofold elevation of troponin-T), aged 18 years and above, who undergo primary percutaneous revascularization (PCI) and have confirmed initial TIMI 0 or 1 in the infarct related coronary artery.

Exclusion Criteria:

* Significant liver disease
* Thrombolytic therapy
* History of prior myocardial infarction
* Current atrial fibrillation
* History of congestive heart failure
* History of migraine headache
* Significant valvular heart disease, primary myocardial disease
* Cardiogenic shock (sRR <90mmHg or need for inotropic support)
* Child-bearing potential
* Inability to read, understand and sign the informed consent
* Life expectancy <3y
* Prior organ transplantation
* Medication with konazoles, ritonavir, rifampicin and sulfonyl-urea derivatives
* Participation in another clinical study
* Metal implants contraindicating CMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion determined by CMR | 3 days

SECONDARY OUTCOMES:
Final infarct size determined by CMR | 3 days
Left ventricular function determined by CMR | 3 days/ 6 months (6-months Remodeling-substudy)
Plasma NT-BNP | 30 days/ 6 months (6-months substudy)
Enzymatic infarct size (CK levels) | 3 days
ECG ST-segment resolution | 1 hour
Markers of inflammation | 24 hours/ 30 days
Major adverse cardiac events (MACE) (cardiovascular death, re-hospitalization for unstable angina and AMI, hospitalization for worsening heart failure) | 30 days
Liver function | 24hours/ 3 days/ 30 days
Event free survival | 6 months (6-months substudy)
Holter ECG | 3 days / 30 days (EP-substudy)

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Lang, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna-Austria, Austria

REFERENCES:
- [Result] Adlbrecht C, Andreas M, Redwan B, Distelmaier K, Mascherbauer J, Kaider A, Wolzt M, Tilea IA, Neunteufl T, Delle-Karth G, Maurer G, Lang IM. Systemic endothelin receptor blockade in ST-segment elevation acute coronary syndrome protects the microvasculature: a randomised pilot study. EuroIntervention. 2012 Apr;7(12):1386-95. doi: 10.4244/EIJV7I12A218. PMID 22522549